CLINICAL TRIAL: NCT02806869
Title: Modernization of in vivo-in Vitro Oral Bioperformance Prediction and Assessment: A Research Study to Evaluate the Performance of an Ibuprofen Oral Dosage Form in the Gastrointestinal Tract of Healthy Adult Volunteers
Brief Title: Modernization of in vivo-in Vitro Oral Bioperformance Prediction and Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Duxin Sun, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FDA_13-RFQ-1116088; HHSF223201310144C (Other Grant/Funding Number: U.S. Food and Drug Administration)
Record Dates: First submitted 2016-05-13; First posted 2016-06-21 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Human Gastrointestinal Physiology Data
MeSH Terms: interventions — Ibuprofen; Tablets

STUDY DESIGN:
Intervention Model Description: This is a parallel study design that allocated subjects into a fasted or fed group. Subject were asked to complete the same study procedures on two occasions.
  Subjects assigned to the fasted or fed group were not crossed-over from one group to the other.

ARMS (2):
- Arm #1 - Fasting State, 2 study visits (Experimental): 1. Single dose of ibuprofen (800 mg tablet) administered with 250 mL of water containing phenol red
  2. Washout period of at least 7 days
  3. Single dose of ibuprofen (800 mg tablet) administered with 250 mL of water containing phenol red
  Interventions: Drug: Single dose of ibuprofen (800 mg tablet)
- Arm #2 - Fed State, 2 study visits (Experimental): 1. Pulmocare, two 8.0 oz (236.6 mL) cans, followed by single dose of ibuprofen (800 mg tablet) administered with 250 mL of water containing phenol red
  2. Washout period of at least 7 days
  3. Pulmocare, two 8.0 oz (236.6 mL) cans, followed by single dose of ibuprofen (800 mg tablet) administered with 250 mL of water containing phenol red
  Interventions: Drug: Single dose of ibuprofen (800 mg tablet); Dietary Supplement: Pulmocare, two 8.0 oz (236.6 mL) cans

INTERVENTIONS:
Drug: Single dose of ibuprofen (800 mg tablet)
Dietary Supplement: Pulmocare, two 8.0 oz (236.6 mL) cans
  Arms: Arm #2 - Fed State, 2 study visits

SUMMARY:
In vivo drug dissolution in the gastrointestinal (GI) tract is largely unmeasured. The purpose of this clinical study was to evaluate the in vivo drug dissolution and systemic absorption of the BCS Class IIa drug ibuprofen under fed and fasted conditions by direct sampling of stomach and small intestinal luminal content. Expanding current knowledge of drug dissolution in vivo will help to establish physiologically relevant in vitro models predictive of drug dissolution.

DETAILED DESCRIPTION:
This is an in vivo study designed to acquire human gastrointestinal (GI) physiology data from healthy subjects under fasting and fed conditions which are necessary for mechanistic absorption model development. Each subject will be asked to complete two GI tube insertion procedures. Subjects will complete this study twice under the same conditions of the GI tract, either fasting state or fed state, in order to provide intra-subject variability. A minimum of 7 days will separate each GI tube insertion procedure. The objectives of this study are, as follows: Objective #1: To acquire human GI physiology data including GI motility, pH of GI fluids, and GI fluid volume under fasting and fed conditions; Objective #2: To measure drug concentration and calculate drug dissolution in the GI tract in vivo under fasting and fed conditions; Objective #3: To monitor plasma drug concentration and evaluate pharmacokinetics of administered drug during GI tube insertion studies under fasting and fed conditions. These in vivo results will be used to validate in vitro dissolution methods and to support computational and mathematical modeling efforts, in order to develop an oral drug product optimization process that may be applied to future drugs to maximize oral drug safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 55.
2. Male or female voluntarily able to give informed consent.

Exclusion Criteria:

1. Adults unable to consent for themselves or mentally incapacitated.
2. Prisoners.
3. Significant clinical illness within 3 weeks prior to Screening.
4. Use of concomitant medications within 2 weeks prior to receiving study drug, including but not limited to prescription drugs, herbal and dietary supplements, over the counter medications, and vitamins. Birth control is permitted.
5. Received an investigational drug within 60 days prior to receiving the study drug.
6. History of gastrointestinal surgery.
7. Surgery within the past 3 months.
8. History of allergy to ibuprofen or other non-steroidal anti-inflammatory drugs (NSAIDs).
9. History of severe allergic diseases including drug allergies, with the exception of seasonal allergies.
10. Any other factor, condition, or disease, including, but not limited to, cardiovascular, renal, hepatic, or gastrointestinal disorders that may, in the opinion of the Investigator, jeopardize the safety of the patient or impact the validity of the study results.
11. History of drug addiction or alcohol abuse within the past 12 months.
12. Pregnant or lactating females.
13. Any clinically significant abnormal lab values during Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01; Primary Completion 2016-11 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duxin Sun, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Yu A, Jackson T, Tsume Y, Koenigsknecht M, Wysocki J, Marciani L, Amidon GL, Frances A, Baker JR, Hasler W, Wen B, Pai A, Sun D. Mechanistic Fluid Transport Model to Estimate Gastrointestinal Fluid Volume and Its Dynamic Change Over Time. AAPS J. 2017 Nov;19(6):1682-1690. doi: 10.1208/s12248-017-0145-x. Epub 2017 Oct 4. PMID 28980204

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (1 Day)
Arm/Group | Arm #1 - Fasting State, 2 Study Visits | Arm #2 - Fed State, 2 Study Visits
Started | 24 | 24
Completed | 13 | 12
Not Completed | 11 | 12
Period: Washout (7 Days)
Arm/Group | Arm #1 - Fasting State, 2 Study Visits | Arm #2 - Fed State, 2 Study Visits
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Arm #1 - Fasting State, 2 Study Visits | Arm #2 - Fed State, 2 Study Visits
Started | 7 | 7
Completed | 7 | 5
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants equals the number of participants who completed the First intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm #1 - Fasting State, 2 Study Visits | Arm #2 - Fed State, 2 Study Visits | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (8.9) | 31.6 (8.8) | 30.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.6 (4.65) | 26.2 (4.61) | 25.9 (4.63)

OUTCOME MEASURES:

1. Primary Outcome: Average Duodenal Fluid pH in Fasted Compared to Fed Participants Administered a Single Dose of Ibuprofen
Description: The pH of duodenal fluid was measured at multiple timepoints over a 7 hour period. The reported value represents the mean and standard deviation of duodenal fluid pH.
Time Frame: from time 0 to 7 hours
Population: Overall Number of Participants Analyzed equals the number of participants who completed the First intervention plus the number of participants who completed the Second Intervention. For Arm #1: Overall Number of Participants Analyzed=13+7=20. For Arm #2: Overall Number of Participants Analyzed=12+5=17.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Arm #1 - Fasting State, 2 Study Visits | Arm #2 - Fed State, 2 Study Visits
Number analyzed (Participants) | 20 | 17
pH | 5.12 (1.64) | 5.36 (1.40)

2. Secondary Outcome: Maximum Duodenal Fluid Concentration of Ibuprofen in Fasted Compared to Fed Participants Administered a Single Dose of Ibuprofen
Description: The concentration of duodenal fluid was measured at multiple timepoints over a 7 hour period. The reported value represents the mean and standard deviation maximum concentration measured in duodenal fluid.
Time Frame: from time 0 to 7 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Arm #1 - Fasting State, 2 Study Visits | Arm #2 - Fed State, 2 Study Visits
Number analyzed (Participants) | 20 | 17
mg/L | 217 (230) | 155 (172)

3. Secondary Outcome: Average Area Under the Plasma Concentration-time Curve (AUC) in Fasted Compared to Fed Participants Administered a Single Dose of Ibuprofen
Description: The plasma concentration of ibuprofen was measured at multiple timepoints over a 24 hour period. The reported value represents the mean and standard deviation of AUC over this time frame.
Time Frame: from time 0 to 24 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*mg/L
Arm/Group | Arm #1 - Fasting State, 2 Study Visits | Arm #2 - Fed State, 2 Study Visits
Number analyzed (Participants) | 20 | 17
h*mg/L | 242 (88.9) | 229 (76.9)

ADVERSE EVENTS:
Arm/Group | Arm #1 - Fasting State, 2 Study Visits | Arm #2 - Fed State, 2 Study Visits
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 1/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm #1 - Fasting State, 2 Study Visits (N=24) | Arm #2 - Fed State, 2 Study Visits (N=24)
hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The variability associated with concentration-time profile in the gastrointestinal tract could not be associated with participant specific factors given the small study sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No